CLINICAL TRIAL: NCT06179966
Title: The Effect of Dance and Massage Applied by Partners at Birth on Birth Pain, Comfort and Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırklareli University (Other)
Responsible Party: Principal Investigator, Ayca Solt Kirca, Asssociate professor, Kırklareli University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KırklareliAS-10
Record Dates: First submitted 2023-12-12; First posted 2023-12-22 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Pain
Keywords: massage; dance; endorphin massage; postpartum comfort
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dance group (Experimental): The application will be taught to the participants' spouses by the researcher after they are admitted to labor, and the spouses will be asked to do it to the participants at regular intervals.
  Interventions: Other: Dance group
- Massage group (Experimental): After admission to travaya, the researcher will teach the pregnant woman's husband practically and the spouses will massage the participants' backs at certain intervals.
  Interventions: Other: Massage group
- Control Group (No Intervention): Routine midwifery care will be provided, and no applications other than routine midwifery care will be performed.

INTERVENTIONS:
Other: Dance group — The application will be taught to the participants' spouses by the researcher after they are admitted to labor, and the spouses will be asked to do it to the participants at regular intervals.
  Arms: Dance group
Other: Massage group — After admission to travaya, the researcher will teach the pregnant woman's husband practically and the spouses will massage the participants' backs at certain intervals.
  Arms: Massage group

SUMMARY:
Pregnancy and the moment of birth are important processes that women will remember throughout their lives and will always leave a mark on their lives. Birth pain is expressed as the most severe pain that women experience throughout their lives (although there is no standard measure due to the combination of different factors). Labor pain; It differs from other types of pain in that it is part of the natural process, occurs within a limited period of time, and the mother willingly endures this pain due to factors such as reuniting with her baby at the end of the process. Due to the possible negative effects of labor pain on maternal and fetal health, the American Society of Anesthesiologists (ASA) and the American Congress of Obstetricians and Gynecologists (ACOG) accept labor pain as an indication that should be treated. recommends that this pain be taken under control. Nowadays, non-pharmacological methods such as "massage, pilates ball, music therapy, acupuncture, aromatherapy" are widely used to manage pain during birth. Massage, which is among the non-pharmacological methods, is the oldest treatment and sensual stimulation method in the world. Massage is generally the first choice method because it has no side effects and is easy to apply. Studies have shown that massage applied during birth provides physical and psychological relief, reduces pain, anxiety, agitation and depressive mood, and increases maternal satisfaction. Determining birth satisfaction is important as it is an indicator of the health status of the mother and newborn as well as the quality of intrapartum care.Birth dance is a combination of music therapy and freedom of movement methods, which is one of the non-pharmacological methods.

Birth dance begins in the active phase of the first stage of labor in order to reduce the pain perceived by the woman and to provide emotional support, and continues until the end of the first stage. The woman is given the opportunity to move rhythmically with someone she prefers (spouse/partner, mother, midwife, etc.), accompanied by relaxing light music. In addition to the music and body movements included in the dance, it is aimed to increase the effectiveness of the applied method by adding spouse/partner support and upright positions and at the same time to provide emotional support to the woman.

DETAILED DESCRIPTION:
Pregnancy and the moment of birth are important processes that women will remember throughout their lives and will always leave a mark on their lives. Birth pain is expressed as the most severe pain that women experience throughout their lives (although there is no standard measure due to the combination of different factors). Labor pain; It differs from other types of pain in that it is part of the natural process, occurs within a limited period of time, and the mother willingly endures this pain due to factors such as reuniting with her baby at the end of the process. Due to the possible negative effects of labor pain on maternal and fetal health, the American Society of Anesthesiologists (ASA) and the American Congress of Obstetricians and Gynecologists (ACOG) accept labor pain as an indication that should be treated. recommends that this pain be taken under control. Different pharmacological and non-pharmacological methods are used to reduce labor pain. Advantages of non-pharmacological methods; These include reducing the rate of use of drugs and eliminating the risk of side effects, being easy and applicable to all individuals, and not imposing an economic burden on the individual.

Nowadays, non-pharmacological methods such as "massage, pilates ball, music therapy, acupuncture, aromatherapy" are widely used to manage pain during birth. Massage, which is among the non-pharmacological methods, is the oldest treatment and sensual stimulation method in the world. Massage is generally the first choice method because it has no side effects and is easy to apply. Studies have shown that massage applied during birth provides physical and psychological relief, reduces pain, anxiety, agitation and depressive mood, and increases maternal satisfaction. Determining birth satisfaction is important as it is an indicator of the health status of the mother and newborn as well as the quality of intrapartum care.

Birth dance is a combination of music therapy and freedom of movement methods, which is one of the non-pharmacological methods.

Birth dance begins in the active phase of the first stage of labor in order to reduce the pain perceived by the woman and to provide emotional support, and continues until the end of the first stage. The woman is given the opportunity to move rhythmically with someone she prefers (spouse/partner, mother, midwife, etc.), accompanied by relaxing light music. In addition to the music and body movements included in the dance, it is aimed to increase the effectiveness of the applied method by adding spouse/partner support and upright positions and at the same time to provide emotional support to the woman.

ELIGIBILITY:
Inclusion Criteria:

* knowing Turkish

  * Being over 18 years old
  * Having a second vaginal birth
  * Being able to go through the labor process with his/her spouse
  * Dilation ≤5cm during vaginal examination during admission to labor
  * Pregnancy period is between 36-40 weeks
  * Agreeing to participate in the research with a voluntary consent form
  * Do not use any non-pharmacological method before admission to labor. not to have used
  * Not using any analgesic or anesthetic medication during labor.

Exclusion Criteria:

* Having any chronic disease (DM, HT, Heart Disease)

  * Receiving psychiatric treatment (Pharmacotherapy and/or Psychotherapy)
  * Presence of a risky pregnancy that prevents normal birth (oligohydramnios, polyhydramnios, twin pregnancy, placental anomalies, presentation and position anomalies)
  * Presence of a wound that disrupts skin integrity
  * Having given birth 3 or more times
  * Being the first pregnancy
  * Exceeding term (>40 weeks) or premature birth (<36 weeks)
  * Presence of previous uterine surgery (caesarean section indication)
  * Not having a partner during labor
  * Have the necessary examination findings to be accepted into the specified research.

not having

* The birth process ends with a cesarean section
* Having an operative birth (vacuum, forceps)
* Wants to leave the research voluntarily.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 105 (Actual)
Dates: Start 2023-03-03 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-05 (Actual)

PRIMARY OUTCOMES:
Introductory Information Form | 1 hour
  sociodemographic characteristics, medical and obstetric pregnancy history, the woman's current pregnancy, prenatal and postpartum period

SECONDARY OUTCOMES:
Visual Comparison Scale | during the birth
  Visual Comparison Scale (VAS = Visual Analog Scale = VAS) is a reliable scale used in children over the age of seven and conscious patients to determine the severity of pain. The patient is asked to mark his/her own pain on a 10-centimeter line with no pain on one end and the worst possible pain on the other end. Evaluation is made by giving points between 0-10. Evaluation of GKS; It is defined as no pain: 0 cm, mild pain: 0.5 cm - 3.0 cm, moderate pain: 3.5 cm - 6.5 cm, severe pain: 7.0 cm - 10.0 cm.
Postpartum Comfort Scale | 6 hours after birth
  WHO; It is a scale that can be used appropriately and safely in measuring the postpartum comfort of mothers who have given birth by normal birth or cesarean section, in meeting postpartum comfort needs, and in evaluating the outcome as a concrete indicator of the outcome. DSKÖ consists of 34 items. A 5-point Likert-type scale scoring system was used to enable an evaluation for each item that determines the situation to be measured. For each item, expressions and scoring ranging from "completely agree" (5 points) to "strongly disagree" (1 point) were made. The lowest score to be obtained from the scale is 34 and the highest score is 170. The average value is determined by dividing the total score obtained from the scale by the number of items and the result is shown in the 1-5 distribution. Basically, low comfort is expressed as 1 and high comfort is expressed as 5.
Person-Centered Maternity Care Scale | 6 hours after birth
  he Turkish form consists of 21 items and 3 sub-dimensions. Except for items 6, 11 and 13 (5 options and coded as 0, 1, 2, 3, 4), the remaining items have 4 options ("no, never" 0, "yes, a few times" 1, "yes, most of the time" "time" is scored as 2, "yes, always" is scored as 3). The lowest score that can be obtained from the total scale is 0, the highest score is 66, the lowest score that can be obtained from the "Valuable and Respectful Care" sub-dimension (2,3,4,5) is 0. The highest score is 12, the lowest score that can be obtained from the sub-dimension "Communication and Autonomy" (1,6,7,8,9,10,11,14) is 0, the highest score is 26, "Supportive Care" (12,13,15,16). The lowest score that can be obtained from the sub-dimension (17,18,19,20,21) is 0 and the highest score is 28. As the score increases, mother-focused care increases
Birth Satisfaction Scale | 2 hours after birth
  DMS consists of 30 Likert-type questions. The score that can be obtained from the scale varies between 30-150 points. As the score obtained from the scale increases, satisfaction with birth increases. Three main themes were identified in the scale: Quality of care (home assessment, birth environment, adequate support and communication with healthcare personnel); personal characteristics of women (ability to cope with childbirth, sense of control, preparation for birth, communication with the baby); Stress experienced during the birth process (difficulty during the birth process, birth injury, perception of receiving adequate medical care, medical interventions, experience of pain, prolonged labor, and the baby's health).

CONTACTS AND LOCATIONS:
Overall Officials: KÜBRA YAVAS, Principal Investigator — TEKIRDAG CORLU STATE HOSPITAL
Locations (1):
- Tekirdag Corlu State Hospital, Tekirdağ, Turkey (Türkiye)